CLINICAL TRIAL: NCT06834061
Title: Added Value of Ultrasonography in the Diagnosis, Management, and Follow-Up of Carpal Tunnel Syndrome
Status: Recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Anas Zahra, Lecturer of Neurosurgery, Faculty of Medicine, KafrElsheikh University, KafrElsheikh, Egypt., Kafrelsheikh University
Other Study IDs: KFSIRB200-513
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Ultrasonography; Diagnosis; Management; Follow-Up; Carpal Tunnel Syndrome
MeSH Terms: conditions — Disease; Carpal Tunnel Syndrome | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound group: All patients underwent high-resolution real-time sonography of the carpal tunnel (both hands) using an Ultrasound (US) machine and a 12 MHz linear array transducer. US examination will be performed before and 3 months after surgery.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — All patients underwent high-resolution real-time sonography of the carpal tunnel (both hands) using an Ultrasound (US) machine and a 12 MHz linear array transducer. US examination will be performed before and 3 months after surgery.

SUMMARY:
This study aims to assess the ultrasound (US) and nerve conduction studies (NCS) as a tool for diagnosis, treatment planning and follow-up of patients with carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is one of the most common upper extremity compression neuropathies and is caused by compression of the median nerve in the carpal tunnel at the wrist.

The ultrasound (US) is a follow-up option as a diagnostic tool in CTS. It is a readily available non-invasive tool which has a shorter examination time. It can measure a number of median nerve parameters, including size, vascularity (using power Doppler) and mobility (using dynamic imaging). In addition,the US provides information on anatomical variations of the median nerve and surrounding structures that may be a causative factor in CTS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Patients with carpal tunnel syndrome.

Exclusion Criteria:

* History of wrist surgery (including carpal tunnel injection) or fracture.
* Clinical or electrophysiological evidence of an accompanying condition that mimics carpal tunnel syndrome or interferes with its evaluation, such as proximal median neuropathy, cervical radiculopathy or polyneuropathy.
* History of underlying disorders associated with carpal tunnel syndrome such as diabetes mellitus, rheumatoid arthritis, pregnancy, acromegaly or hypothyroidism.
* Electrodiagnostic findings suggestive of co-existing neurological disorders.
* Subclinical sensory polyneuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will be carried out on 60 patients with CTS admitted in KafrElsheikh University Hospitals over a period of 6 months starting from approval of the Medical Sciences Ethics Committee of KafrElsheikh Faculty of Medicine and all the included patients will provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ultrasound in diagnosis of carpal tunnel syndrome | Intraoperatively
  Sensitivity of ultrasound in diagnosis of carpal tunnel syndrome will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.